CLINICAL TRIAL: NCT02381795
Title: An Open Label, Pilot Study Evaluating the Efficacy and Safety of the Use of Nasal Carbon Dioxide for the Treatment of Episodic Cluster Headache
Brief Title: Pilot Study Evaluating the Use of Nasal Carbon Dioxide for the Treatment of Cluster Headache
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated at the request of the financial sponsor.
Sponsor: Cady, Roger, M.D. (Individual)
Collaborators: Capnia, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-001CA
Record Dates: First submitted 2015-03-03; First posted 2015-03-06 (Estimated); Results first posted 2018-05-01 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-07

CONDITIONS: Cluster Headache
MeSH Terms: conditions — Cluster Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nasal Carbon Dioxide (Experimental): 0.17 liters (L) of carbon dioxide (CO2) will be delivered through two 10 second administrations in each nostril, up to 6 times, to treat one attack (total of 1.0 L CO2). Subjects may treat up to three cluster headache attacks during the treatment phase of this study (total of 3.0 L (CO2).
  Interventions: Drug: Nasal Carbon Dioxide

INTERVENTIONS:
Drug: Nasal Carbon Dioxide

SUMMARY:
This is an open label, investigator-sponsored, pilot study. Subjects agreeing to participate in the study and meeting the eligibility criteria assessed at the screening visit will be enrolled in the study. The length of time between screening and treatment will last between 0 days to a maximum of 12 weeks. Subjects who enter the screening phase during a cluster headache episode and meet the study eligibility criteria can immediately enter the treatment phase and may opt to treat their cluster headache episode in the clinic. Subjects who are not in a cluster headache episode, who meet initial screening eligibility criteria, can remain in the screening phase for up to 12 weeks until their next cluster episode begins. Upon initiation of a cluster headache episode, subjects will enter the treatment period. Subjects will be trained on the proper use of the hand-held dispenser containing carbon dioxide (CO2 )calibrated to deliver 0.5 standard liters per minute (SLPM). This dispenser will be provided for use in the clinic or home. Subjects will be instructed to use the nasal CO2 dispenser, 10 seconds/nostril, as needed up to 6 times to treat one attack. Each dose must be separated by 3-5 minutes. Subjects should treat only one attack in a 24-hour period. Subjects may treat up to three cluster headache attacks during the treatment phase of this study. One hour after the first dose, subjects can choose to treat with investigator-approved rescue medication. Subjects will be asked to complete an online diary after the completion of the dosing. Diary assessments will collect pain severity, nasal CO2 usage, acute medication usage, satisfaction of treatment, number of cluster attacks, and unusual symptoms. Subjects will be contacted by phone within 3 days of the first use of the nasal CO2 dispenser to assess adverse events (AEs) and medication usage. A total of 25 subjects will enter the treatment period and be instructed to treat up to 3 cluster headaches with nasal CO2. Within 7 days of treating their last cluster headache episode, subjects will return for an end of study visit.

ELIGIBILITY:
Inclusion Criteria:

* Male and female, 18 years of age and older.
* History of episodic cluster headache, as defined by International Classification of Headache Disorders (ICHD), third edition, beta version guidelines (ICHD-3 beta, Cephalalgia 2013).
* History of cluster headache attack-free remission periods lasting > 1 month within the previous year.
* Stable on medications, including those for the treatment of cluster headache prevention/prophylaxis, for at least 60 days prior to baseline (including, but not limited to, verapamil, lithium, melatonin, any anticonvulsant, any systemic corticosteroid or steroid injection, occipital nerve block, other cranial or extracranial nerve block, or any neurostimulation treatment).

Note: Subjects are allowed to use their usual standard of care for the acute/abortive treatment of acute cluster attacks 60 or more minutes after the initial dose, limited to the following: triptans; high-flow oxygen.

* If female and of childbearing potential, have a negative urine pregnancy test at the time of Screening.

  a. To not be considered childbearing potential a subject must be surgically sterile, have had a hysterectomy or tubal ligation, post-menopausal for at least 1 year, or otherwise incapable of pregnancy.
* Capable of completing online headache diary with access to internet.
* Able to provide written Informed Consent.

Exclusion Criteria:

* Recent nasal/midface trauma (< 3 months)
* Recent nasal/sinus surgery (< 3 months).
* Severe respiratory distress in the last 6 months.
* Neoplasm such as Angiofibroma, sinus tumor, granuloma.
* Nasal congestion present more than 10 days with fever (temperature ≥ 100.4 °F) and nasal mucous is an abnormal color.
* Surgery to treat cluster headache.
* History of aneurysm, intracranial hemorrhage, brain tumors or significant head trauma.
* Structural intracranial or cervical vascular lesions that may potentially cause headache attacks.
* Other significant pain problems (including cancer pain, fibromyalgia, and trigeminal neuralgia) that might confound the study assessments in the investigator opinion.
* Psychiatric disorder, which in the opinion of the Investigator, may interfere with the study.
* Pregnant, actively trying to become pregnant, or breastfeeding, and/or is unwilling to use an accepted form of birth control.
* Skin around and inside the nasal passage that is dry, cracked, oozing, or bleeding.
* Recurrent nose bleeds, which in the opinion of the Investigator, may interfere with the study.
* Is participating in any other therapeutic clinical investigation or has participated in a clinical trial and received treatment in the preceding 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-07; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinvest/A Division of Banyan Group, Inc., Springfield, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Nasal Carbon Dioxide: 0.17 liters (L) of carbon dioxide (CO2) will be delivered through two 10 second administrations in each nostril, up to 6 times, to treat one attack (total of 1.0 L CO2). Subjects may treat up to three cluster headache attacks during the treatment phase of this study (total of 3.0 L (CO2).
  Nasal Carbon Dioxide
Period: Overall Study
Arm/Group | Nasal Carbon Dioxide
Started | 10
Completed | 7
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Study Terminated | 2

BASELINE CHARACTERISTICS:
Arm/Group | Nasal Carbon Dioxide
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (13.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Headache Pain Intensity
Description: Greatest change in headache pain intensity post treatment (at any time point within 30 minutes of Nasal CO2 administration) - pre-treatment. Pain intensity will be measured as follows: 0 = no pain, 1 = mild pain, 2 = moderate pain, and 3 = severe pain. Full Range values were calculated change values, and do not represent the full range of the scale.
Time Frame: Immediately preceeding treatment to 30 minutes post-treatment
Population: Enrolled subjects reporting at least one headache during study period. One enrolled subject did not experience any headaches during the study period and thus was not included in the analysis.
Measure: Mean (Full Range); unit: units on a scale
Units Other Than Participants: Cluster Headaches
Arm/Group | Nasal Carbon Dioxide
Number analyzed (Participants) | 9
Number analyzed (Cluster Headaches) | 23
units on a scale | -0.826 [-3 to 1]

ADVERSE EVENTS:
Time Frame: 25 weeks
Arm/Group | Nasal Carbon Dioxide
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 5/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nasal Carbon Dioxide (N=10)
Cluster headache (Nervous system disorders) | 1 (1)
Goitre (Endocrine disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Lacrimation increase (Eye disorders) | 2 (4)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-28): https://cdn.clinicaltrials.gov/large-docs/95/NCT02381795/Prot_SAP_000.pdf